CLINICAL TRIAL: NCT00005580
Title: Phase I Study of Bryostatin 1 (NSC 339555) and Fludarabine in Patients With Chronic Lymphocytic Leukemia and Indolent Non-Hodgkin's Lymphoma
Brief Title: Bryostatin + Fludarabine in Treating Patients With Chronic Lymphocytic Leukemia or Relapsed Indolent Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: National Cancer Institute
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066433; P30CA016059 (NIH); MCV-CCHR-9801-2C; NCI-T97-0116
Record Dates: First submitted 2000-05-02; First posted 2003-01-27 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2010-02

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent cutaneous T-cell non-Hodgkin lymphoma; Waldenstrom macroglobulinemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; refractory chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; B-cell chronic lymphocytic leukemia; refractory hairy cell leukemia; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult T-cell leukemia/lymphoma; prolymphocytic leukemia; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, T-Cell, Cutaneous; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — bryostatin 1; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: bryostatin 1
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase I trial to study the effectiveness of bryostatin 1 plus fludarabine in treating patients who have chronic lymphocytic leukemia or relapsed, indolent non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxic effects and maximum tolerated dose of bryostatin 1 and fludarabine in patients with symptomatic or advanced chronic lymphocytic leukemia or relapsed indolent non-Hodgkin's lymphoma.
* Monitor apoptosis, differentiation, and protein kinase C activity in leukemic lymphocytes exposed in vivo to bryostatin 1 and fludarabine.
* Observe the antitumor activity of this combination therapy in these patients.

OUTLINE: This is a dose-escalation, multicenter study. Patients are assigned to one of two treatment groups.

* Group I: Patients receive bryostatin 1 IV over 24 hours followed by fludarabine IV over 30 minutes daily on days 1-5.
* Group II: Patients receive fludarabine IV over 30 minutes daily on days 1-5 followed by bryostatin 1 IV over 24 hours.

In both groups, courses repeat every 4 weeks for patients with stable or responding disease.

Cohorts of 3-6 patients receive escalating doses of fludarabine and bryostatin 1 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity. Once the MTD for fludarabine is determined, the dose of bryostatin 1 is escalated.

PROJECTED ACCRUAL: Approximately 30-60 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed chronic lymphocytic leukemia

  * Stage I (symptomatic or with bulky lymphadenopathy)
  * Stage II, III, or IV
  * Prior chemotherapy allowed, including fludarabine or other purine nucleoside analog therapy OR
* Histologically confirmed indolent non-Hodgkin's lymphoma

  * Progressive or relapsed following chemotherapy
* Includes the following histologies:

  * B-cell chronic lymphocytic leukemia/prolymphocytic leukemia/lymphomas

    * Lymphoplasmacytoid lymphoma (Waldenstrom's)/immunocytoma
    * Mantle cell lymphoma
    * Follicular lymphoma

      * Small cell
      * Mixed small and large cell
      * Diffuse (predominately small cell type)
    * Marginal zone B-cell lymphoma

      * Extranodal (MALT-type with or without monocytoid B-cells)
      * Provisional subtype: nodal (with or without monocytoid B-cells)
    * Provisional entity: splenic marginal zone lymphoma (with or without villous lymphocytes)
    * Hairy cell leukemia
* Peripheral T-cell and NK-cell neoplasms

  * T-cell chronic lymphocytic leukemia/polylymphocytic leukemia
  * Large granular lymphocyte leukemia

    * T-cell type
    * NK-cell type
  * Mycosis fungoides/Sezary's syndrome (cutaneous T-cell lymphoma)
* No CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,000/mm3
* Platelet count at least 75,000/mm3
* Hemoglobin at least 8 g/dL
* Coombs negative

Hepatic:

* AST/ALT no greater than 2.5 times upper limit of normal
* Bilirubin no greater than 2 mg/mL

Renal:

* Creatinine clearance at least 40 mL/min

Other:

* No concurrent neurologic condition
* No other concurrent medical condition that would preclude study
* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 3 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No concurrent systemic immunoglobulin therapy
* No prior bone marrow or peripheral stem cell transplantation

Chemotherapy:

* See Disease Characteristics
* At least 3 weeks since prior systemic chemotherapy

Endocrine therapy:

* No concurrent systemic glucocorticoid therapy

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1998-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grant, MD, Study Chair — Massey Cancer Center
Locations (3):
- United States (3):
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Result] Roberts JD, Smith MR, Feldman EJ, Cragg L, Millenson MM, Roboz GJ, Honeycutt C, Thune R, Padavic-Shaller K, Carter WH, Ramakrishnan V, Murgo AJ, Grant S. Phase I study of bryostatin 1 and fludarabine in patients with chronic lymphocytic leukemia and indolent (non-Hodgkin's) lymphoma. Clin Cancer Res. 2006 Oct 1;12(19):5809-16. doi: 10.1158/1078-0432.CCR-05-2730. PMID 17020988